CLINICAL TRIAL: NCT04124276
Title: Evaluation of Efficacy of Lycium Barbarum Polysaccharide in Patients With Major Depressive Disorder: a Randomized,Placebo-controled Trial
Brief Title: Evaluation of Efficacy of Lycium Barbarum Polysaccharide in Patients With Major Depressive Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Psychiatric Hospital (Other Government)
Collaborators: Fifth Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Kangguang Lin, Deputy director, Department of Affective Disorder, Guangzhou Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Guangzhou Brain LBPMD
Record Dates: First submitted 2019-10-05; First posted 2019-10-11 (Actual); Last update posted 2020-10-30 (Actual); Status verified 2020-10

CONDITIONS: Major Depressive Disorder; Depression; Depressive Disorder
Keywords: Major Depressive Disorder; Lycium barbarum polysaccharide
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Depressive Disorder | interventions — lycium barbarum polysaccharide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lycium barbarum polysaccharide (Experimental): Experimental group takes Lycium barbarum polysaccharide (LBP) tablet (300mg/day) for 6 weeks
  Interventions: Dietary Supplement: Lycium barbarum polysaccharide
- Placebo (Placebo Comparator): Placebo control group takes placebo (300mg/day) for 6 weeks. The placebos are the same with the LBP tablets in appearance and taste.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lycium barbarum polysaccharide — Experimental groups take Lycium barbarum polysaccharide (LBP) (300mg/day) for 6 weeks
  Arms: Lycium barbarum polysaccharide
Dietary Supplement: Placebo — Placebo control group takes placebo (300mg/day) for 6 weeks.
  Arms: Placebo

SUMMARY:
Lycium barbarum, a traditional Chinese herbal medicine, is a commonly used herb in the traditional Chinese pharmacopoeia. Its main active ingredient, lycium barbarum polysaccharide (LBP), is reported to have neuroprotective effects. Animal studies suggested that LBP has neuroprotective effect on optic ganglion cells. In animal models of depression, LBP can improve depressive symptom by improving synaptic plasticity. However, its clinical effect remains to be studied. We will conduct a 6-week double-blind, randomized, placebo-con-trolled trial in patients with major depressive disorder (MDD). The purpose of this clinical trial is to investigate the efficacy of LBP in patients with MDD.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-60 years old
2. Sex: both men and women
3. Compliance with the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5) diagnostic criteria for major depressive disorder
4. Hamilton Depression Scale scored more than 18 points.
5. No contraindication of taking Lycium barbarum polysaccharide

Exclusion Criteria:

1. Comorbidity with other mental disorders
2. Severe somatic diseases
3. Current use of traditional Chinese medicine
4. Suicide concept, attempt, act and attempted suicide
5. Psychiatric symptoms
6. Taking hormones and endocrine drugs
7. Long-term use of wolfberry in recent three months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 284 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Reduction rate of Hamilton Depression Scale (HDRS) | 4weeks, 6weeks
  HDRS is used to measure the depressive severity；its measured time range is within the past week. In this study, version of 24-items is used. The patients are depressed when the total score are greater than 19 points, and there are no depression when the total scores are less than points. Clinical control, HDRS score reduction rate≥75%; significant progress, 50%≤HDRS score reduction rate < 75%; progress, 25%≤HDRS score reduction rate < 50%; ineffectiveness, HDRS score reduction rate < 25%. significant efficiency = (clinical control + significant progress) / sample number×100%.

SECONDARY OUTCOMES:
Changes in depressive severity measured by Beck Depression Inventory (BDI) scale and Kessler Scale(K10) | 4 weeks, 6 weeks
  BDI scale is used to measure depressive severity by patients themselves. It's made of 21 items. Circle the number in front of the sentence that best suits your situation in according to the feeling for a week. The total score is obtained by adding up the delimited scores of each item. There is depression when the total score is greater than 15 points and there is no depression when the total score is less than 10 points. The K10 is a widely used, simple self-report measure of psychological distress which can be used to identify those in need of further assessment of depression and anxiety
Changes in sleep quality | 4 weeks, 6 weeks
  Changes in Pittsburgh Sleep Quality Index (PSQI) scale. PSQI scale is used to evaluate sleep quality for last month. It's made of 7 items; every item is scored 1-4 point. Total score is obtained by adding up the points of 7 items. Total score range is 0~21 point. The sleep quality is worse when the total score is higher.
Changes in cognitive function | 4 weeks, 6 weeks
  Cognitive function is assessed using the THINC-it. The THINC-it was recently developed by the THINC-it Task Force (http://thinc.progress.im/en) with the principal goal of time-efficient screening of cognitive impairments specifically among individuals with major depressive disorder as a routine component of their clinical care. THINC-it is a digitized cognitive assessment battery comprised of carefully selected gamified variations of well-known cognitive tasks (Spotter [Choice Reaction Time], Symbol Check [One-Back], Codebreaker [Digit Symbol Substitution Test], Trails [Trail Making Test-Part B]), and the Perceived Deficits Questionnaire for Depression-5-item (PDQ-5-D), a subjective self-report scale.
Changes in social adaptive levels | 4 weeks, 6 weeks
  Measured by Global Assessment Function (GAF) scale. GAF scale is used to evaluate the condition and social adaptability in psychiatry patients. It's divided into 1 to 100 grades. The lower the score, the more serious the disease is. 91-100 points shows that the patients have good social adaptation and normal mental status.
Changes in serum brain-derived neurotrophic factor (BDNF) levels | 6 weeks
  We measure the serum BDNF levels by enzyme linked immunosorbent assay (ELISA)
Changes in serum triglyceride levels | 6 weeks
  The blood of patients are sent to clinical laboratory of our hospital to measure serum triglyceride levels
Changes in serum total cholesterol levels | 6 weeks
  The blood of patients are sent to clinical laboratory of our hospital to measure serum total cholesterol levels

CONTACTS AND LOCATIONS:
Overall Officials: Kangguang Lin, MD, PhD, Principal Investigator — Guangzhou Brain Hospital (Guangzhou Huiai Hospital)
Locations (1):
- Guangzhou Brain Hospital (Guangzhou Huiai Hospital), Guanzhou, Guangdong, China